CLINICAL TRIAL: NCT05539378
Title: Biomarkers of Brain Clearance During Sleep
Brief Title: Exploring the Link Between Sleep and Brain Clearance
Acronym: BBCDS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital, Zurich (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: BBCDS
Record Dates: First submitted 2022-07-20; First posted 2022-09-14 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Healthy Aging
MeSH Terms: interventions — Acoustic Stimulation; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (participant and outcomes assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auditory Stimulation (Experimental): Auditory Stimulation during sleep
  Interventions: Behavioral: Auditory Stimulation
- No Auditory Stimulation (Sham Comparator): Playing no tones during sleep but still recording brain activity
  Interventions: Behavioral: Sham (no stimulation)

INTERVENTIONS:
Behavioral: Auditory Stimulation — enhancement of sleep slow wave activity through acoustic stimulation
  Arms: Auditory Stimulation
Behavioral: Sham (no stimulation) — Playing no tones during sleep but still recording brain activity
  Arms: No Auditory Stimulation

SUMMARY:
The purpose of this study is to assess the link between sleep and the clearance of waste products from the brain. This will be assessed in a group of healthy older adults.

DETAILED DESCRIPTION:
First, the investigators want to assess the relationship between sleep parameters and markers for brain clearance, assessed with MRI and blood samples. Second, the investigators want to probe whether associations can be influenced by modulation of sleep parameters by means of auditory stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Participation in previous longitudinal cohort studies at the study site
* Ability to provide written and verbal informed consent
* Fluency in the German language
* Stable home situation that allows for reliable application of the intervention for the duration of the study
* Ability to apply the intervention for the duration of the study, either alone or with support from a co-habitant
* For women: Hormonal contraception, if menstrual cycle is still present or has been present within a year
* Good general health status, normal cognitive function

Exclusion Criteria:

* Failure or inability to give informed consent
* Inability to follow the procedures of the investigation
* For women: pregnancy or breastfeeding
* Presence of sleep disorders (e.g. sleep apnoea, narcolepsy, restless leg syndrome, insomnia, rapid eye movement (REM) sleep disorder)
* Shift-work or a home situation that requires several awakenings during the night (e.g. newborn)
* History of serious illness likely to interfere with study outcomes
* Presence or history of a diagnosed neuropsychiatric illness
* Current diagnosis of uncontrolled or poorly controlled diabetes
* Current cancer of the brain or unstable cancer undergoing treatment
* Evidence of serious atherosclerotic cardiovascular disease

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Correlation between EEG slow wave activity (uV) and cerebrospinal fluid flow (ml/min) from phase contrast MRI | 2 weeks
Correlation between EEG slow wave activity (uV) and diffusivity (mm2/s) from diffusion MRI | 2 weeks
Correlation between EEG slow wave activity (uV) and perfusion (ml/min/100 ml) from arterial spin labelling MRI | 2 weeks
Correlation between EEG slow wave activity (uV) and beta-amyloid (pg/ml) | 2 weeks
Correlation between EEG slow wave activity (uV) and tau (pg/ml) | 2 weeks

SECONDARY OUTCOMES:
Correlation between EEG slow wave activity (uV) and fatigue, assessed via the fatigue severity scale (FSS) questionnaire | 2 weeks
Correlation between EEG slow wave activity (uV) and sleepiness, assessed with the Epworth Sleepiness Scale questionnaire | 2 weeks
Correlation between EEG slow wave activity (uV) and memory function, assessed with the Hopkins Verbal Learning Test (memory score) | 2 weeks
Correlation between EEG slow wave activity (uV) and attention, assessed with the Trail Making Test (time to completion) | 2 weeks
Correlation between EEG slow wave activity (uV) and C-Reactive Protein (mg/L), assessed from a blood sample | 2 weeks
Correlation between EEG slow wave activity (uV) and TNF-alpha (pg/L), assessed from a blood sample | 2 weeks
Correlation between EEG slow wave activity (uV) and interleukins (pg/L), assessed from a blood sample | 2 weeks
Correlation between EEG slow wave activity (uV) and executive function (summary score, dimensionless) | 2 weeks
Correlation between EEG slow wave activity (uV) and neuro-metabolite levels (mmol) from magnetic resonance spectroscopy | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anton Gietl, Principal Investigator — Institute for Regenerative Medicine, University of Zurich
Locations (1):
- Institute for Regenerative Medicine, University Hospital Zurich, Zurich, Switzerland